CLINICAL TRIAL: NCT04407494
Title: Diagnostic Value of Patient - Reported and Clinically Verified Olfactory Disorders in a Population Tested for COVID-19
Brief Title: Diagnostic Value of Patient - Reported and Clinically Verified Olfactory Disorders (COVID-19)
Acronym: COVID-OLFA
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0176
Record Dates: First submitted 2020-05-27; First posted 2020-05-29 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; COVID-19; Diagnostic value; Sensitivity; Specificity; Prevalence; Positive predictive value; Negative predictive value; Epidemiology; Diagnostic test; Anosmia; Ageusia; Olfactory disorders; Gustatory disorders; Smell disorders; Taste disorders
MeSH Terms: conditions — COVID-19; Hypersensitivity; Anosmia; Ageusia; Olfaction Disorders; Taste Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — NC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19: Healthcare workers and adult outpatients attending the COVID-19 screening center of the University Hospital of Montpellier, France.
  Interventions: Biological: Reporting of anosmia, ageusia and other clinical symptoms

INTERVENTIONS:
Biological: Reporting of anosmia, ageusia and other clinical symptoms — Reporting of anosmia, ageusia and other clinical symptoms related to COVID-19 - CODA test - SARS-CoV2 RT-PCR and ELISA

SUMMARY:
Participants are healthcare workers and adult outpatients referred in a COVID-19 screening center. Patients-reported symptoms are collected, then participants underwent a simple olfactory test (CODA for Clinical Olfactory Dysfunction Assessment), prior to swabbing for SARS-CoV-2 diagnosis (RT-PCR). We aimed to evaluate the prevalence of smell and taste disorders, and to calculate the diagnostic value of patient-reported and clinically verified smell disorders in persons with suspected COVID-19.

ELIGIBILITY:
Inclusion criteria:

* Symptoms compatible with COVID-19
* Close exposure to a confirmed COVID-19 index case
* Ambulatory (asymptomatic, or if symptomatic, did not require hospitalisation, thus with initial mild disease)

Exclusion criteria:

* known history of smell and taste disorders
* testing inability (cognitive impairment, non native French speakers, test malingering)
* testing contraindication (children, pregnancy, breastfeeding, specific allergies).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthcare workers and adult outpatients attending the COVID-19 screening center of the University Hospital of Montpellier, France.
Sampling Method: Probability Sample
Enrollment: 809 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic values of anosmia and ageusia for COVID-19 | at inclusion
  Diagnostic values of anosmia and ageusia for COVID-19 with questionnaire

SECONDARY OUTCOMES:
Diagnostic values of CODA | at inclusion
  Diagnostic values of CODA (Clinical Olfactory dysfunction Assessment) score for COVID-19 : Simple, fast, semi-objective olfactory test developed for epidemic context

CONTACTS AND LOCATIONS:
Overall Officials: Fréderic VENAIL, PU-PH, Study Director — UH Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC